CLINICAL TRIAL: NCT00614900
Title: Prevalence and Influence of Pulmonary Hypertension in COPD Patients
Brief Title: Prevalence of Pulmonary Hypertension in COPD Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Andersen, MD, University of Aarhus
Other Study IDs: PreKPH-08; jnr 2007-0206
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: COPD; pulmonary hypertension; NT-proBNP; 6 minutes walk test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of an increased pulmonary blood pressure amongst patients with chronic obstructive pulmonary disease (COPD)is unclear. So is the impact of abnormal pulmonary blood pressure on symptoms. The aim of this study is to determine the prevalence of an increased pulmonary blood pressure in 200 patients with COPD. Furthermore we will investigate if lung function test results and blood tests can predict an increased pulmonary blood pressure, and explore whether COPD patients with a high pulmonary blood pressure have more symptoms that their co-patients.

DETAILED DESCRIPTION:
The prevalence of pulmonary hypertension in patients with chronic obstructive pulmonary disease (COPD) is unclear. The presence of an abnormally increased pulmonary blood pressure worsens the prognosis of COPD, but the patients are not currently diagnosed or treated for pulmonary hypertension. The aim of this study is to determine the prevalence of pulmonary hypertension in 200 patients with COPD and explore whether it worsens functional capacity and symptoms. Furthermore we will look into whether blood gas values, NT-proBNP, CRP and lung function test result can predict which patients are at risk of having pulmonary hypertension.

Methods: All patients will be screened by echocardiography. Those with signs of pulmonary hypertension will be admitted to right heart catheterization for direct measurements of pulmonary haemodynamics.

All patients will perform a 6 minutes walk test and spirometry. Blood levels of NT-proBNP and CRP will be measured. Life quality by the St. George Questionnaire and contacts to the health care system is also assessed. Differences in these parameters are analyzed among patients with no, moderate or severe pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Prior admittance to hospital with exacerbation in COPD
* Informed consent

Exclusion Criteria:

* Exacerbation in COPD less than 6 weeks before examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients have been admitted to hospital with an exacerbation in COPD in 2006.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hilberg, Md, Dr.med., Study Director — Aarhus Universitetshospital, Aarhus Sygehus
Locations (1):
- Department of pulmonary diseases, Aarhus Sygehus, Aarhus, Denmark